CLINICAL TRIAL: NCT02119156
Title: An Open-label, Non-randomized, 52-Week Study to Evaluate Treatment Holidays and Rebound Phenomenon After Treatment With Belimumab 10 mg/kg in Systemic Lupus Erythematosus Subjects
Brief Title: Belimumab Treatment Holiday and Treatment Re-start Study in Lupus Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 116027
Expanded Access: NCT03125486 (No longer available)
Record Dates: First submitted 2014-04-17; First posted 2014-04-21 (Estimated); Results first posted 2020-01-31 (Actual); Last update posted 2020-01-31 (Actual); Status verified 2020-01

CONDITIONS: Systemic Lupus Erythematosus
Keywords: treatment holiday; PGA; belimumab; Lymphostat-B; rebound; SELENA SLEDAI; Systemic Lupus Erythematosus; immunogenicity
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — belimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Treatment Holiday Group (Experimental): Subjects in the Treatment Holiday Group will undergo a 6 month belimumab treatment holiday while remaining on standard of care SLE therapy, then re-start belimumab therapy for 6 months while receiving standard of care SLE therapy.
  Interventions: Drug: Belimumab
- Control Group (Active Comparator): Subjects in the Control Group will continue to receive monthly belimumab therapy, in addition to standard of care SLE therapy for 52 weeks.
  Interventions: Drug: Belimumab
- Long-Term Discontinuation Group (No Intervention): Subjects in the Long-Term Discontinuation Group have elected to discontinue further belimumab therapy and will remain on standard of care SLE therapy as directed by the investigator, and agree to return for monthly visits for 52 weeks.

INTERVENTIONS:
Drug: Belimumab — Monthly intravenous infusions dosed as 10 mg/kg body weight
  Arms: Control Group; Treatment Holiday Group

SUMMARY:
This study will assess the effect of a 24-week withdrawal followed by a 28-week reintroduction of belimumab 10 mg/kg plus standard of care medications in subjects with stable low systemic lupus erythematosus (SLE) disease activity. Rebound phenomenon will be assessed for subjects who have permanently withdrawn from further belimumab treatment.

DETAILED DESCRIPTION:
This study will assess the effect of a 24-week withdrawal of belimumab followed by a 28-week reintroduction of belimumab 10 mg/kg plus standard of care medications on immunogenicity, markers of biological activity, efficacy, and safety in subjects with stable low systemic lupus erythematosus (SLE) disease activity. Additionally, this study will assess rebound phenomenon in subjects with any disease level of SLE who have permanently withdrawn from further belimumab treatment

ELIGIBILITY:
Inclusion Criteria:

* Received a minimun of 6 months therapy with with belimumab 10 mg/kg in their current SLE belimumab continuation study.
* Be 18 years of age at the Day 0 visit.
* Non-prenant, non-lactating females willing to comply with specific birth control requirements as set forth in the protocol.
* Able to provide written informed consent to participate.
* Subjects who wish to enroll in the control group and the group taking a 6 month belimumab treatment holiday will need a SELENA SLEDAI score of 3 or less after the minimum of 6 months belimumab therapy, as well as having C3 and C4 complement levels at or above the lower limit of the central laboratory reference range, and are on a stable SLE treatment regimen during the 30 day screening period prior to Day 0.
* Subjects who wish to enroll in the long-term discontinuation group have voluntarily withdrawn from their continuation studies.

Exclusion Criteria:

* Subjects who have developed clinical evidence of significant, unstable or uncontrolled, acute or chronic diseases not due to SLE, or experienced an adverse event (AE) in their belimumab continuation study that could, in the opinion of the principle investigator, put the subject at undue risk.
* Subjects who have developed any other medical diseases, laboratory abnormalities, or conditions that, in the opinion of the principle investigator, makes the subject unsuitable for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2014-05-13 (Actual); Primary Completion 2018-12-14 (Actual); Study Completion 2018-12-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (16):
- United States (3):
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Manhasset, New York
  - GSK Investigational Site, Dallas, Texas
- China (4):
  - GSK Investigational Site, Hefei, Anhui
  - GSK Investigational Site, Suzhou, Jiangsu
  - GSK Investigational Site, Hangzhou, Zhejiang
  - GSK Investigational Site, Beijing
- Japan (6):
  - GSK Investigational Site, Chiba
  - GSK Investigational Site, Ehime
  - GSK Investigational Site, Hokkaido
  - GSK Investigational Site, Miyagi
  - GSK Investigational Site, Nagasaki
  - GSK Investigational Site, Tokyo
- South Korea (3):
  - GSK Investigational Site, Daegu
  - GSK Investigational Site, Seoul
  - GSK Investigational Site, Suwon, Kyonggi-do

REFERENCES:
- [Derived] Bae SC, Bass DL, Chu M, Curtis P, Dimelow R, Harvey L, Ji B, Kurrasch R, Muzaffar S, Punwaney R, Roth DA, Song YW, Xie W, Zhang F. The effect of 24-week belimumab treatment withdrawal followed by treatment restart in patients with SLE: an open-label, non-randomised 52-week study. Arthritis Res Ther. 2022 Feb 16;24(1):46. doi: 10.1186/s13075-022-02723-y. PMID 35172878

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was multi-center study to evaluate temporary discontinuation of belimumab 10 milligram(mg)/kilogram(kg) for 24 weeks followed by reintroduction of belimumab 10 mg/kg Intravenous (IV) for 28 weeks, in participants with low Systemic Lupus Erythematosus (SLE) disease activity receiving belimumab plus standard of care.
Pre-assignment Details: A total of 80 participants were enrolled for this study. Participants were enrolled across 20 sites in China, Japan, Korea and the United States.
Groups:
- Long-term Discontinuation Group: Participants in this group discontinued belimumab 10 mg/kg therapy for 52 weeks but remained on standard of care therapy. Participants from BEL114333 (NCT01597622), BEL112233 (NCT00724867) and BEL112626 (NCT00583362) were part of this group. Participants had been treated with belimumab for at least 6 months in one of these continuation studies but had withdrawn from belimumab therapy for no longer than 8 weeks prior to entry into this study.
- Treatment Control Group: Participants in this group continued to receive monthly belimumab 10 mg/kg therapy, in addition to standard of care SLE therapy for 52 weeks. Participants from BEL113750 (NCT01345253) and BEL114333 (NCT01597622) were part of this group. Participants had been treated with belimumab for at least 6 months in one of these continuation studies prior to entry into this study. Eligible participants on completion of 52-weeks entered Maintenance period and received belimumab 10 mg/kg every 4 weeks until Week 48 of subsequent years (Maintenance is Year 2, 3, 4).
- Treatment Holiday Group: Participants in the Treatment Holiday Group underwent a 24-week belimumab treatment holiday while remaining on standard of care SLE therapy, then re-started belimumab therapy for further 28 weeks while receiving standard of care SLE therapy. Participants from BEL113750 (NCT01345253) and BEL114333 (NCT01597622) were part of this group. Participants had been treated with belimumab for at least 6 months in one of these continuation studies prior to entry into this study. Eligible participants on completion of 52-weeks entered Maintenance period and received belimumab 10 mg/kg every 4 weeks until Week 48 of subsequent years (Maintenance is Year 2, 3, 4).
Period: Treatment Phase (Up to 52 Weeks)
Arm/Group | Long-term Discontinuation Group | Treatment Control Group | Treatment Holiday Group
Started | 39 | 29 | 12
Completed | 33 | 27 | 11
Not Completed | 6 | 2 | 1
Not completed — Study Terminated By Sponsor | 0 | 0 | 1
Not completed — Withdrawal by Subject | 4 | 0 | 0
Not completed — Protocol Violation | 1 | 2 | 0
Not completed — Physician Decision | 1 | 0 | 0
Period: Maintenance (Up to 48 Weeks of Year 2-4)
Arm/Group | Long-term Discontinuation Group | Treatment Control Group | Treatment Holiday Group
Started | 0 (Long-term discontinuation participants were not allowed in Maintenance period) | 16 (Eligible participants of Treatment control and holiday group on completion of 52-weeks were included) | 10 (Eligible participants of Treatment control and holiday group on completion of 52-weeks were included)
Completed | 0 | 6 | 3
Not Completed | 0 | 10 | 7
Not completed — Study Terminated By Sponsor | 0 | 10 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Long-term Discontinuation Group | Treatment Control Group | Treatment Holiday Group | Total
Number analyzed (Participants) | 39 | 29 | 12 | 80
Age, Continuous [Mean (Standard Deviation); unit: Years] | 38.9 (12.01) | 40.6 (9.76) | 38.1 (8.04) | 39.4 (10.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 27 | 9 | 71
  Male | 4 | 2 | 3 | 9
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White/Caucasian/European Heritage | 9 | 0 | 0 | 9
  Asian: Central/South Asian Heritage | 1 | 0 | 0 | 1
  Asian: East Asian Heritage | 23 | 27 | 4 | 54
  Asian: Japanese Heritage | 0 | 2 | 8 | 10
  African American/African Heritage | 5 | 0 | 0 | 5
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Median Time to First SLE Flare Index (SFI)
Description: SFI Flare was defined as a mild/moderate or severe flare according to the modified Safety of Estrogen in Lupus National Assessment Systemic Lupus Erythematosus Disease Activity Index (SELENA SLEDAI) SLE Flare Index (modified excluded severe flares from the SELENA SLEDAI flare assessment that were triggered only by an increase in SELENA SLEDAI score to >12).Time to first SFI flare is defined as the number of days from Day 0 visit date to the date the participant has a flare (event date - Day 0 visit date + 1) in the 52 Week/Holiday phase; (event date - treatment re-start date + 1) in the Re-start Holiday phase. Day 0 visit date is defined as Day 0 from present study. Median time to first SFI flare is reported; estimated using the product-limit method.
Time Frame: Up to 52 weeks
Population: Intent-to-Treat (ITT) Population comprised of all participants who enrolled in the study, excluding screen failures.
Measure: Median (Inter-Quartile Range); unit: Days
Groups:
- Treatment Holiday Group - Holiday Phase: Participants in the Treatment Holiday Group underwent a 24-week belimumab treatment holiday while remaining on standard of care SLE therapy, Holiday Phase was Day 0 visit to Week 24/Treatment Re-start phase. Participants from BEL113750 (NCT01345253) and BEL114333 (NCT01597622) were part of this group. Participants had been treated with belimumab for at least 6 months in one of these continuation studies prior to entry into this study. In the event of a severe flare, participants were allowed to enter Maintenance Phase and receive belimumab 10 mg/Kg every 4 weeks until Week 48 of subsequent years (Maintenance is Year 2, 3, 4).
- Treatment Holiday Group - Re-start Phase: Following Treatment holiday phase for 24 weeks, participants re-started belimumab therapy for 28 weeks while receiving standard of care SLE therapy for 52 weeks. Re-start Phase started one day after Week 24 up to Week 52. Participants from BEL113750 (NCT01345253) and BEL114333 (NCT01597622) were part of this group. Participants had been treated with belimumab for at least 6 months in one of these continuation studies prior to entry into this study. Eligible participants on completion of 52-weeks entered Maintenance period and received belimumab 10 mg/kg every 4 weeks until Week 48 of subsequent years (Maintenance is Year 2, 3, 4).
Arm/Group | Long-term Discontinuation Group | Treatment Control Group | Treatment Holiday Group - Holiday Phase | Treatment Holiday Group - Re-start Phase
Number analyzed (Participants) | 39 | 29 | 12 | 11
Days | 183.0 [91.0 to 370.0] | NA [365.0 to NA] — NA indicates that "Due to low event rates of participants in treatment groups, the median time and/or interquartile range could not be estimated" | NA [30.0 to NA] — NA indicates that "Due to low event rates of participants in treatment groups, the median time and/or interquartile range could not be estimated" | NA [NA to NA] — NA indicates that "Due to low event rates of participants in treatment groups, the median time and/or interquartile range could not be estimated"

2. Secondary Outcome: Rate of SLE Index Flare Per Subject Year
Description: Rate per subject year of SFI flare was calculated as total number of flares divided by total subject years in interval. The total subject years for each participant was calculated as (Week 52/ Exit visit date minus Day 0 visit date + 1) for Long-term discontinuation and treatment control groups. For treatment holiday phase group the subject-years for each participant was calculated as (Week 24/Treatment Re-start/Exit visit date minus Day 0 Visit date + 1)/365.25. For re-start treatment holiday phase group the subject-years for each participant was calculated as (Week 52/Exit visit date minus Week 24/Treatment Re-start date + 1)/365.25. Day 0 visit date is defined as Day 0 from present study.
Time Frame: Up to 52 weeks
Population: ITT Population
Measure: Number; unit: Flares per Subject-year
Arm/Group | Long-term Discontinuation Group | Treatment Control Group | Treatment Holiday Group - Holiday Phase | Treatment Holiday Group - Re-start Phase
Number analyzed (Participants) | 39 | 29 | 12 | 11
Flares per Subject-year | 2.1 | 0.6 | 1.0 | 0.3

3. Secondary Outcome: Median Time to First Severe SFI Flare
Description: The SLE Flare Index categorizes SLE flare as "mild or moderate" or "severe" based on a positive assessment for at least 1 of 5 variables as follows: Change in SELENA SLEDAI score from the most recent assessment to current; Change in signs or symptoms of disease activity; Change in prednisone dosage; Use of new medications for disease activity or hospitalization; Change in Physician's Global Assessment (PGA) score; Hospitalization for SLE activity is an additional category included only for a severe flare. Time to first severe flare is defined as (event date-Day 0 visit date) + 1 for Long-term discontinuation, treatment control groups and holiday phase group. For holiday phase group data censored at last flare assessment by treatment re-start date. Time to first severe flare is defined as (event date-treatment re-start date) + 1 for Re-start treatment holiday group. Median time to first severe SFI flare is reported; estimated using the product-limit method.
Time Frame: Up to 52 weeks
Population: ITT Population.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Long-term Discontinuation Group | Treatment Control Group | Treatment Holiday Group - Holiday Phase | Treatment Holiday Group - Re-start Phase
Number analyzed (Participants) | 39 | 29 | 12 | 11
Days | NA [327.0 to NA] — NA indicates that "Due to low event rates of participants in treatment groups, the median time and/or interquartile range could not be estimated" | NA [NA to NA] — NA indicates that "Due to low event rates of participants in treatment groups, the median time and/or interquartile range could not be estimated" | NA [NA to NA] — NA indicates that "Due to low event rates of participants in treatment groups, the median time and/or interquartile range could not be estimated" | NA [NA to NA] — NA indicates that "Due to low event rates of participants in treatment groups, the median time and/or interquartile range could not be estimated"

4. Secondary Outcome: Number of Participants With Evidence of Rebound
Description: Rebound is defined as SELENA SLEDAI score during the first 24 weeks that exceeds the Baseline SELENA SLEDAI score in the participant's respective original parent study. Baseline is defined as the Day 0 visit from the parent study. SELENA SLEDAI assessments consist of 24 individual weighted items in which signs and symptoms, laboratory tests, and physician's assessment for each of 9 organ systems are given a weighted score and summed if present (marked 'Yes') at the time of the visit or in the preceding 10 days. The maximum theoretical score is 105 (all 24 descriptors present simultaneously) with 0 indicating inactive disease (marked 'No'). Any time during the first 24 weeks of this study has been reported.
Time Frame: Up to 24 weeks
Population: ITT Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Long-term Discontinuation Group | Treatment Control Group | Treatment Holiday Group
Number analyzed (Participants) | 39 | 29 | 12
Participants | 2 | 2 | 0

5. Secondary Outcome: Number of Participants With Confirmed True Positive Belimumab Anti-drug Antibodies (ADA)
Description: Immunogenicity assay results were categorized as negative or positive. A persistent positive result was defined as a positive post-Day 0 visit immunogenic response that occurred for at least 2 consecutive assessments or a single result at the final assessment. A transient positive result was defined as a single post-Day 0 visit positive immunogenic response that did not occur at the final assessment. Any time post-Day 0 visit data are reported (or post-Week 24 for Treatment Holiday - Restart phase). Day 0 visit date is defined as Day 0 from present study.
Time Frame: Up to 52 weeks
Population: ITT Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Long-term Discontinuation Group | Treatment Control Group | Treatment Holiday Group - Holiday Phase | Treatment Holiday Group - Re-start Phase
Number analyzed (Participants) | 39 | 29 | 12 | 11
Participants
  Negative | 39 | 29 | 12 | 11
  Persistent positive | 0 | 0 | 0 | 0
  Transient positive | 0 | 0 | 0 | 0

6. Secondary Outcome: Percentage Change From Baseline in Immunoglobulin
Description: Serum samples were collected at indicated time-points for analysis of immunoglobulins: Immunoglobulin G (IgG), Immunoglobulin A (IgA), and Immunoglobulin M (IgM). Baseline is defined as the Day 0 visit from parent studies. Percentage change from Baseline is equal to 100* (value at specified visit minus Baseline value) divided by Baseline value.
Time Frame: Baseline (Day 0 from parent studies); Day 0 and 8, 16, 24, 32, 40, 48 and 52 weeks
Population: ITT Population. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | Long-term Discontinuation Group | Treatment Control Group | Treatment Holiday Group - Holiday Phase | Treatment Holiday Group - Re-start Phase
Number analyzed (Participants) | 39 | 29 | 12 | 11
Percent change
  IgA,Day 0,n=31,29, 12,0: number analyzed (Participants) | 31 | 29 | 12 | 0
  IgA,Day 0,n=31,29, 12,0 | -19.205 [-38.406 to -7.229] | -25.909 [-35.168 to -16.901] | -22.193 [-33.468 to -14.278] |
  IgA,Week 8,n=37,29, 11,0: number analyzed (Participants) | 37 | 29 | 11 | 0
  IgA,Week 8,n=37,29, 11,0 | -21.028 [-41.897 to -11.066] | -31.455 [-37.166 to -24.186] | -24.242 [-36.981 to -14.213] |
  IgA, Week 16,n=36,27, 11,0: number analyzed (Participants) | 36 | 27 | 11 | 0
  IgA, Week 16,n=36,27, 11,0 | -22.052 [-39.715 to -8.880] | -31.016 [-36.676 to -23.432] | -20.202 [-38.381 to -4.975] |
  IgA, Week 24,n=31,27, 11,0: number analyzed (Participants) | 31 | 27 | 11 | 0
  IgA, Week 24,n=31,27, 11,0 | -20.570 [-34.101 to 3.271] | -28.000 [-34.097 to -21.033] | -21.711 [-35.533 to 5.240] |
  IgA, Week 32,n=34,27,0,10: number analyzed (Participants) | 34 | 27 | 0 | 10
  IgA, Week 32,n=34,27,0,10 | -11.243 [-29.004 to 3.004] | -29.703 [-37.615 to -19.697] |  | -23.363 [-39.164 to -1.875]
  IgA, Week 40,n=33,25,0,11: number analyzed (Participants) | 33 | 25 | 0 | 11
  IgA, Week 40,n=33,25,0,11 | -10.769 [-33.575 to 2.715] | -30.617 [-37.143 to -26.934] |  | -24.579 [-33.891 to 1.990]
  IgA, Week 48,n=33,27,0,10: number analyzed (Participants) | 33 | 27 | 0 | 10
  IgA, Week 48,n=33,27,0,10 | -16.000 [-27.848 to 10.850] | -34.091 [-37.867 to -19.767] |  | -33.936 [-42.105 to 6.883]
  IgA, Week 52,n=33,27,0,10: number analyzed (Participants) | 33 | 27 | 0 | 10
  IgA, Week 52,n=33,27,0,10 | -14.859 [-28.646 to 9.346] | -30.698 [-38.806 to -17.128] |  | -31.663 [-40.102 to 0.498]
  IgG,Day 0,n=39,29, 12,0: number analyzed (Participants) | 39 | 29 | 12 | 0
  IgG,Day 0,n=39,29, 12,0 | -13.939 [-35.349 to 3.571] | -29.524 [-35.645 to -14.872] | -19.481 [-33.330 to -9.757] |
  IgG,Week 8,n=37,29, 11,0: number analyzed (Participants) | 37 | 29 | 11 | 0
  IgG,Week 8,n=37,29, 11,0 | -19.169 [-37.209 to -0.877] | -29.048 [-35.795 to -6.897] | -25.571 [-31.788 to -16.234] |
  IgG, Week 16,n=36,27, 11,0: number analyzed (Participants) | 36 | 27 | 11 | 0
  IgG, Week 16,n=36,27, 11,0 | -16.169 [-37.881 to 8.306] | -29.818 [-35.714 to -5.172] | -21.642 [-29.870 to -18.721] |
  IgG, Week 24,n=31,27, 11,0: number analyzed (Participants) | 31 | 27 | 11 | 0
  IgG, Week 24,n=31,27, 11,0 | -17.982 [-34.545 to 0.662] | -26.241 [-32.571 to -7.080] | -17.886 [-26.623 to -8.955] |
  IgG, Week 32,n=34,27,0,10: number analyzed (Participants) | 34 | 27 | 0 | 10
  IgG, Week 32,n=34,27,0,10 | -9.798 [-34.146 to 3.653] | -23.288 [-34.220 to -8.420] |  | -18.611 [-24.725 to -9.459]
  IgG, Week 40,n=34,25,0,11: number analyzed (Participants) | 34 | 25 | 0 | 11
  IgG, Week 40,n=34,25,0,11 | -6.955 [-36.842 to 4.878] | -25.532 [-34.286 to -15.575] |  | -26.484 [-27.473 to -16.418]
  IgG, Week 48,n=33,27,0,10: number analyzed (Participants) | 33 | 27 | 0 | 10
  IgG, Week 48,n=33,27,0,10 | -14.063 [-34.082 to 2.222] | -25.133 [-33.945 to -6.897] |  | -20.596 [-29.870 to -8.209]
  IgG, Week 52,n=33,27,0,10: number analyzed (Participants) | 33 | 27 | 0 | 10
  IgG, Week 52,n=33,27,0,10 | -11.258 [-34.457 to 9.756] | -23.596 [-29.655 to -14.359] |  | -23.754 [-25.974 to -18.543]
  IgM,Day 0,n=31,29, 12,0: number analyzed (Participants) | 31 | 29 | 12 | 0
  IgM,Day 0,n=31,29, 12,0 | -47.059 [-67.333 to -26.761] | -53.608 [-64.583 to -41.463] | -44.326 [-63.895 to -25.516] |
  IgM,Week 8,n=37,29, 11,0: number analyzed (Participants) | 37 | 29 | 11 | 0
  IgM,Week 8,n=37,29, 11,0 | -49.174 [-65.672 to -34.868] | -53.659 [-64.583 to -46.262] | -50.943 [-70.621 to -31.325] |
  IgM, Week 16,n=36,27, 11,0: number analyzed (Participants) | 36 | 27 | 11 | 0
  IgM, Week 16,n=36,27, 11,0 | -50.077 [-61.922 to -30.099] | -54.945 [-61.224 to -43.103] | -45.926 [-70.690 to -19.277] |
  IgM, Week 24,n=31,27, 11,0: number analyzed (Participants) | 31 | 27 | 11 | 0
  IgM, Week 24,n=31,27, 11,0 | -39.496 [-53.153 to -36.184] | -50.909 [-62.963 to -34.483] | -45.161 [-65.517 to -8.511] |
  IgM, Week 32,n=34,27,0,10: number analyzed (Participants) | 34 | 27 | 0 | 10
  IgM, Week 32,n=34,27,0,10 | -34.887 [-48.936 to -18.000] | -52.577 [-66.667 to -31.250] |  | -46.548 [-56.863 to -12.766]
  IgM, Week 40,n=34,25,0,11: number analyzed (Participants) | 34 | 25 | 0 | 11
  IgM, Week 40,n=34,25,0,11 | -37.870 [-46.847 to -20.667] | -52.381 [-65.556 to -41.304] |  | -48.889 [-67.241 to -10.638]
  IgM, Week 48,n=33,27,0,10: number analyzed (Participants) | 33 | 27 | 0 | 10
  IgM, Week 48,n=33,27,0,10 | -31.707 [-54.667 to -11.765] | -53.636 [-63.333 to -40.625] |  | -48.268 [-58.824 to -14.458]
  IgM, Week 52,n=33,27,0,10: number analyzed (Participants) | 33 | 27 | 0 | 10
  IgM, Week 52,n=33,27,0,10 | -30.921 [-53.750 to -4.348] | -51.648 [-67.532 to -46.429] |  | -57.966 [-72.414 to -30.120]

7. Secondary Outcome: Percentage Change From Baseline in Autoantibody:Anti-double Stranded Deoxyribonucleic Acid (dsDNA)
Description: Blood samples were collected at indicated time-points for analysis of autoantibodies like dsDNA. Baseline is defined as the Day 0 visit from parent studies. Percentage change from Baseline is equal to 100* (Value at specified visit minus Baseline value) divided by Baseline value.
Time Frame: Baseline (Day 0 from parent studies); Day 0 and 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48 and 52 weeks
Population: as for outcome 6
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | Long-term Discontinuation Group | Treatment Control Group | Treatment Holiday Group - Holiday Phase | Treatment Holiday Group - Re-start Phase
Number analyzed (Participants) | 39 | 29 | 12 | 11
Percent change
  Day 0,n=39,29,12, 0: number analyzed (Participants) | 39 | 29 | 12 | 0
  Day 0,n=39,29,12, 0 | -82.8 [-90.3 to -38.5] | -69.4 [-88.7 to -46.2] | -81.3 [-84.9 to -52.0] |
  Week 4,n=39,29,12, 0: number analyzed (Participants) | 39 | 29 | 12 | 0
  Week 4,n=39,29,12, 0 | -82.8 [-92.2 to -46.1] | -65.9 [-89.0 to -53.8] | -83.2 [-90.0 to -51.6] |
  Week 8,n=37,29, 11,0: number analyzed (Participants) | 37 | 29 | 11 | 0
  Week 8,n=37,29, 11,0 | -74.3 [-89.5 to -33.7] | -70.3 [-89.5 to -47.5] | -81.6 [-87.7 to -54.5] |
  Week 12,n=38,29, 11,0: number analyzed (Participants) | 38 | 29 | 11 | 0
  Week 12,n=38,29, 11,0 | -77.3 [-89.1 to -28.2] | -68.9 [-90.1 to -50.0] | -85.0 [-88.6 to -53.0] |
  Week 16,n=36,27, 11,0: number analyzed (Participants) | 36 | 27 | 11 | 0
  Week 16,n=36,27, 11,0 | -78.4 [-89.7 to -33.9] | -72.8 [-91.2 to -34.1] | -79.7 [-86.4 to -64.1] |
  Week 20,n=34,27, 11,0: number analyzed (Participants) | 34 | 27 | 11 | 0
  Week 20,n=34,27, 11,0 | -82.8 [-90.3 to -33.7] | -70.3 [-91.9 to -50.0] | -79.9 [-88.3 to -55.2] |
  Week 24,n=31,27, 11,0: number analyzed (Participants) | 31 | 27 | 11 | 0
  Week 24,n=31,27, 11,0 | -82.8 [-92.6 to -41.2] | -71.8 [-91.9 to -38.5] | -75.0 [-87.4 to -54.5] |
  Week 28,n=35,27,0,10: number analyzed (Participants) | 35 | 27 | 0 | 10
  Week 28,n=35,27,0,10 | -69.8 [-88.9 to -28.1] | -72.3 [-91.9 to -46.2] |  | -79.9 [-88.3 to -56.8]
  Week 32,n=34,27,0,11: number analyzed (Participants) | 34 | 27 | 0 | 11
  Week 32,n=34,27,0,11 | -77.9 [-90.0 to -33.3] | -71.4 [-89.5 to -50.0] |  | -79.6 [-91.3 to -57.1]
  Week 36,n=34,27,0,11: number analyzed (Participants) | 34 | 27 | 0 | 11
  Week 36,n=34,27,0,11 | -75.1 [-88.4 to -13.5] | -71.0 [-92.9 to -50.0] |  | -80.8 [-90.8 to -62.9]
  Week 40,n=34,25,0,11: number analyzed (Participants) | 34 | 25 | 0 | 11
  Week 40,n=34,25,0,11 | -73.6 [-91.2 to -4.8] | -87.4 [-93.7 to -70.2] |  | -79.9 [-90.1 to -53.2]
  Week 44,n=34,27,0,10: number analyzed (Participants) | 34 | 27 | 0 | 10
  Week 44,n=34,27,0,10 | -62.0 [-90.3 to -21.4] | -77.7 [-94.0 to -52.3] |  | -82.5 [-91.1 to -50.0]
  Week 48,n=33,27,0,10: number analyzed (Participants) | 33 | 27 | 0 | 10
  Week 48,n=33,27,0,10 | -71.8 [-90.3 to -21.4] | -76.6 [-92.8 to -50.0] |  | -80.6 [-86.4 to -63.3]
  Week 52,n=33,27,0,10: number analyzed (Participants) | 33 | 27 | 0 | 10
  Week 52,n=33,27,0,10 | -65.3 [-91.7 to -15.9] | -78.3 [-91.5 to -38.5] |  | -79.5 [-91.1 to -64.3]

8. Secondary Outcome: Percentage Change From Baseline in Autoantibody: Antinuclear Antibody (ANA)
Description: Blood samples were collected at indicated time-points for analysis of autoantibodies like ANA. Only participants who had an ANA value measured in INDEX at the parent studies Baseline were included in this analysis. Baseline is defined as the Day 0 visit from parent studies. Percentage change from Baseline is equal to 100* (Value at specified visit minus Baseline value) divided by Baseline value.
Time Frame: Baseline (Day 0 from parent studies); Day 0 and 24 and 52 weeks
Population: as for outcome 6
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | Long-term Discontinuation Group | Treatment Control Group | Treatment Holiday Group - Holiday Phase | Treatment Holiday Group - Re-start Phase
Number analyzed (Participants) | 21 | 27 | 10 | 9
Percent change
  Day 0,n=21,27, 10,0: number analyzed (Participants) | 21 | 27 | 10 | 0
  Day 0,n=21,27, 10,0 | -15.044 [-29.716 to 4.193] | -24.938 [-58.221 to 0.000] | -32.336 [-47.741 to -26.843] |
  Week 24,n=20,26, 10,0: number analyzed (Participants) | 20 | 26 | 10 | 0
  Week 24,n=20,26, 10,0 | 5.723 [-9.113 to 24.347] | -27.434 [-62.747 to 0.000] | -29.771 [-44.978 to -13.643] |
  Week 52,n=19,26,0,9: number analyzed (Participants) | 19 | 26 | 0 | 9
  Week 52,n=19,26,0,9 | -16.455 [-56.522 to 21.800] | -45.961 [-66.917 to -11.765] |  | -35.539 [-43.928 to -20.586]

9. Secondary Outcome: Percentage Change From Baseline in Complement Levels
Description: Blood samples were collected at indicated time-points for analysis of complement levels like complement 3 (C3) and complement 4 (C4). Baseline is defined as the Day 0 visit from parent studies. Percentage change from Baseline is equal to 100* (Value at specified visit minus Baseline value) divided by Baseline value.
Time Frame: Baseline (Day 0 from parent studies); Day 0 and 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48 and 52 weeks
Population: as for outcome 6
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | Long-term Discontinuation Group | Treatment Control Group | Treatment Holiday Group - Holiday Phase | Treatment Holiday Group - Re-start Phase
Number analyzed (Participants) | 39 | 29 | 12 | 11
Percent change
  C3, Day 0,n=39,27,12, 0: number analyzed (Participants) | 39 | 27 | 12 | 0
  C3, Day 0,n=39,27,12, 0 | 10.3 [-4.5 to 42.9] | 7.2 [-6.8 to 35.8] | 32.1 [23.7 to 61.5] |
  C3, Week 4,n=39,29,12, 0: number analyzed (Participants) | 39 | 29 | 12 | 0
  C3, Week 4,n=39,29,12, 0 | 15.4 [-2.2 to 42.0] | 16.0 [-7.3 to 27.5] | 14.8 [-6.8 to 46.1] |
  C3,Week 8,n=37,29, 11,0: number analyzed (Participants) | 37 | 29 | 11 | 0
  C3,Week 8,n=37,29, 11,0 | 13.6 [4.3 to 38.3] | 19.8 [-1.0 to 40.6] | 31.4 [17.2 to 60.9] |
  C3,Week 12,n=38,29, 11,0: number analyzed (Participants) | 38 | 29 | 11 | 0
  C3,Week 12,n=38,29, 11,0 | 10.9 [-6.3 to 50.0] | 14.1 [5.2 to 39.1] | 30.4 [24.7 to 75.0] |
  C3,Week 16,n=36,27, 11,0: number analyzed (Participants) | 36 | 27 | 11 | 0
  C3,Week 16,n=36,27, 11,0 | 15.2 [-0.6 to 59.1] | 20.5 [0.0 to 46.7] | 32.2 [20.0 to 62.5] |
  C3,Week 20,n=34,27, 11,0: number analyzed (Participants) | 34 | 27 | 11 | 0
  C3,Week 20,n=34,27, 11,0 | 15.4 [-4.7 to 40.3] | 13.6 [-4.3 to 26.6] | 30.0 [18.3 to 70.3] |
  C3,Week 24,n=31,27, 11,0: number analyzed (Participants) | 31 | 27 | 11 | 0
  C3,Week 24,n=31,27, 11,0 | 17.3 [-7.0 to 41.0] | 19.8 [-1.3 to 58.9] | 44.2 [5.7 to 53.2] |
  C3,Week 28,n=35,27,0,10: number analyzed (Participants) | 35 | 27 | 0 | 10
  C3,Week 28,n=35,27,0,10 | 15.8 [-10.0 to 36.4] | 15.4 [7.8 to 42.2] |  | 31.3 [12.6 to 57.7]
  C3,Week 32,n=34,27,0,11: number analyzed (Participants) | 34 | 27 | 0 | 11
  C3,Week 32,n=34,27,0,11 | 13.8 [0.0 to 53.7] | 21.6 [6.7 to 50.7] |  | 31.6 [16.0 to 69.2]
  C3,Week 36,n=34,27,0,11: number analyzed (Participants) | 34 | 27 | 0 | 11
  C3,Week 36,n=34,27,0,11 | 9.4 [-2.9 to 44.8] | 17.0 [-8.1 to 35.1] |  | 26.0 [11.7 to 67.3]
  C3,Week 40,n=34,25,0,11: number analyzed (Participants) | 34 | 25 | 0 | 11
  C3,Week 40,n=34,25,0,11 | 12.8 [-2.5 to 28.3] | 17.3 [3.1 to 39.7] |  | 41.8 [12.8 to 62.5]
  C3,Week 44,n=34,27,0,10: number analyzed (Participants) | 34 | 27 | 0 | 10
  C3,Week 44,n=34,27,0,10 | 14.1 [0.0 to 29.7] | 22.7 [-6.3 to 51.6] |  | 38.9 [23.0 to 75.0]
  C3,Week 48,n=33,27,0,10: number analyzed (Participants) | 33 | 27 | 0 | 10
  C3,Week 48,n=33,27,0,10 | 15.4 [-5.1 to 35.0] | 15.9 [-4.5 to 41.5] |  | 30.4 [13.8 to 82.7]
  C3,Week 52,n=33,27,0,10: number analyzed (Participants) | 33 | 27 | 0 | 10
  C3,Week 52,n=33,27,0,10 | 5.9 [-9.1 to 25.9] | 21.9 [3.5 to 32.8] |  | 36.5 [7.1 to 77.3]
  C4, Day 0,n=39,27,12, 0: number analyzed (Participants) | 39 | 27 | 12 | 0
  C4, Day 0,n=39,27,12, 0 | 36.4 [-6.3 to 100.0] | 27.8 [11.1 to 128.6] | 70.8 [25.2 to 154.2] |
  C4, Week 4,n=39,29,12, 0: number analyzed (Participants) | 39 | 29 | 12 | 0
  C4, Week 4,n=39,29,12, 0 | 31.6 [10.0 to 100.0] | 47.4 [0.0 to 87.5] | 39.7 [6.7 to 110.4] |
  C4,Week 8,n=37,29, 11,0: number analyzed (Participants) | 37 | 29 | 11 | 0
  C4,Week 8,n=37,29, 11,0 | 37.5 [2.6 to 83.3] | 71.4 [11.8 to 105.6] | 58.3 [33.3 to 183.3] |
  C4,Week 12,n=38,29, 11,0: number analyzed (Participants) | 38 | 29 | 11 | 0
  C4,Week 12,n=38,29, 11,0 | 27.6 [4.5 to 122.2] | 68.4 [12.0 to 121.4] | 64.3 [16.7 to 200.0] |
  C4,Week 16,n=36,27, 11,0: number analyzed (Participants) | 36 | 27 | 11 | 0
  C4,Week 16,n=36,27, 11,0 | 35.4 [13.1 to 158.3] | 50.0 [17.4 to 114.3] | 41.7 [25.0 to 150.0] |
  C4,Week 20,n=34,27, 11,0: number analyzed (Participants) | 34 | 27 | 11 | 0
  C4,Week 20,n=34,27, 11,0 | 32.6 [4.2 to 114.3] | 64.3 [0.0 to 109.1] | 58.3 [17.6 to 166.7] |
  C4,Week 24,n=31,27, 11,0: number analyzed (Participants) | 31 | 27 | 11 | 0
  C4,Week 24,n=31,27, 11,0 | 34.8 [0.0 to 128.6] | 57.1 [15.8 to 125.0] | 66.7 [26.3 to 83.3] |
  C4,Week 28,n=35,27,0,10: number analyzed (Participants) | 35 | 27 | 0 | 10
  C4,Week 28,n=35,27,0,10 | 31.3 [0.0 to 100.0] | 66.7 [8.0 to 100.0] |  | 50.6 [8.3 to 166.7]
  C4,Week 32,n=34,27,0,11: number analyzed (Participants) | 34 | 27 | 0 | 11
  C4,Week 32,n=34,27,0,11 | 27.6 [0.0 to 106.7] | 92.9 [21.7 to 128.6] |  | 58.3 [21.1 to 175.0]
  C4,Week 36,n=34,27,0,11: number analyzed (Participants) | 34 | 27 | 0 | 11
  C4,Week 36,n=34,27,0,11 | 29.2 [0.0 to 100.0] | 50.0 [11.1 to 116.7] |  | 58.3 [25.0 to 183.3]
  C4,Week 40,n=34,25,0,11: number analyzed (Participants) | 34 | 25 | 0 | 11
  C4,Week 40,n=34,25,0,11 | 32.1 [0.0 to 73.3] | 73.3 [29.4 to 112.5] |  | 58.3 [21.1 to 116.7]
  C4,Week 44,n=34,27,0,10: number analyzed (Participants) | 34 | 27 | 0 | 10
  C4,Week 44,n=34,27,0,10 | 20.5 [0.0 to 68.8] | 57.1 [12.0 to 116.7] |  | 60.7 [36.8 to 150.0]
  C4,Week 48,n=33,27,0,10: number analyzed (Participants) | 33 | 27 | 0 | 10
  C4,Week 48,n=33,27,0,10 | 31.3 [-5.9 to 60.0] | 64.3 [15.8 to 114.3] |  | 34.5 [10.5 to 100.0]
  C4,Week 52,n=33,27,0,10: number analyzed (Participants) | 33 | 27 | 0 | 10
  C4,Week 52,n=33,27,0,10 | 17.6 [-5.9 to 62.5] | 63.2 [-4.0 to 126.7] |  | 58.3 [0.0 to 133.3]

10. Secondary Outcome: Percentage Change From Baseline in B Cell Subsets
Description: Blood samples were collected at indicated time-points for analysis of Activated B cells subsets like Activated CD19+CD20+CD69+, cluster of differentiation 20+ (CD20+), Memory CD19+CD20+CD27+, Naive CD19+CD20+CD27-, Plasma CD19+CD20-CD138+, Plasmacytoid CD19+CD20+CD138+, and SLE Subset CD19+CD38b+CD27b+Lymph. Baseline is defined as the Day 0 visit from parent studies. Percentage change from Baseline is equal to 100* (Value at specified visit minus Baseline value) divided by Baseline value.
Time Frame: Baseline (Day 0 from parent studies); Day 0 and 8, 16, 24, 32, 40 and 52 weeks
Population: as for outcome 6
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | Long-term Discontinuation Group | Treatment Control Group | Treatment Holiday Group - Holiday Phase | Treatment Holiday Group - Re-start Phase
Number analyzed (Participants) | 16 | 2 | 8 | 7
Percent change
  Memory CD19+CD20+CD27+, Day 0,n=16,2,8,0: number analyzed (Participants) | 16 | 2 | 8 | 0
  Memory CD19+CD20+CD27+, Day 0,n=16,2,8,0 | -69.0 [-80.9 to -58.9] | -76.1 [-80.0 to -72.2] | -43.2 [-55.0 to 68.3] |
  Memory CD19+CD20+CD27+, Week 8,n=15,2,5,0: number analyzed (Participants) | 15 | 2 | 5 | 0
  Memory CD19+CD20+CD27+, Week 8,n=15,2,5,0 | -73.7 [-85.0 to -60.0] | -78.9 [-80.0 to -77.8] | -50.0 [-71.4 to 50.0] |
  Memory CD19+CD20+CD27+,Week16,n=14,2,6,0: number analyzed (Participants) | 14 | 2 | 6 | 0
  Memory CD19+CD20+CD27+,Week16,n=14,2,6,0 | -83.4 [-93.2 to -66.7] | -69.2 [-80.0 to -58.3] | -60.7 [-80.0 to 0.0] |
  Memory CD19+CD20+CD27+,Week24,n=13,2,6,0: number analyzed (Participants) | 13 | 2 | 6 | 0
  Memory CD19+CD20+CD27+,Week24,n=13,2,6,0 | -86.7 [-93.3 to -78.3] | -59.7 [-69.4 to -50.0] | -65.0 [-71.4 to 0.0] |
  Memory CD19+CD20+CD27+,Week32,n=12,2,0,7: number analyzed (Participants) | 12 | 2 | 0 | 7
  Memory CD19+CD20+CD27+,Week32,n=12,2,0,7 | -85.8 [-91.4 to -72.5] | -73.3 [-80.0 to -66.7] |  | -20.0 [-52.0 to 133.3]
  Memory CD19+CD20+CD27+,Week40,n=13,2,0,7: number analyzed (Participants) | 13 | 2 | 0 | 7
  Memory CD19+CD20+CD27+,Week40,n=13,2,0,7 | -80.0 [-84.2 to -73.9] | -65.6 [-70.0 to -61.1] |  | 0.0 [-48.0 to 83.3]
  Memory CD19+CD20+CD27+,Week52,n=13,2,0,6: number analyzed (Participants) | 13 | 2 | 0 | 6
  Memory CD19+CD20+CD27+,Week52,n=13,2,0,6 | -81.8 [-86.7 to -65.2] | -78.9 [-80.0 to -77.8] |  | -10.0 [-57.1 to 83.3]
  Naive CD19+CD20+CD27-,Day 0,n=16,2,8,0: number analyzed (Participants) | 16 | 2 | 8 | 0
  Naive CD19+CD20+CD27-,Day 0,n=16,2,8,0 | -78.3 [-90.0 to -63.7] | -91.6 [-96.9 to -86.3] | -81.0 [-91.2 to -27.0] |
  Naive CD19+CD20+CD27-,Week 8,n=15,2,5,0: number analyzed (Participants) | 15 | 2 | 5 | 0
  Naive CD19+CD20+CD27-,Week 8,n=15,2,5,0 | -80.5 [-90.4 to -60.0] | -94.3 [-96.5 to -92.2] | -83.0 [-84.6 to -16.7] |
  Naive CD19+CD20+CD27-,Week16,n=14,2,6,0: number analyzed (Participants) | 14 | 2 | 6 | 0
  Naive CD19+CD20+CD27-,Week16,n=14,2,6,0 | -76.4 [-89.9 to -58.1] | -89.6 [-96.9 to -82.4] | -81.0 [-92.3 to -10.6] |
  Naive CD19+CD20+CD27-,Week 24,n=13,2,6,0: number analyzed (Participants) | 13 | 2 | 6 | 0
  Naive CD19+CD20+CD27-,Week 24,n=13,2,6,0 | -45.7 [-90.3 to 38.1] | -92.9 [-95.6 to -90.2] | -54.2 [-71.4 to 34.8] |
  Naive CD19+CD20+CD27-,Week 32,n=12,2,0,7: number analyzed (Participants) | 12 | 2 | 0 | 7
  Naive CD19+CD20+CD27-,Week 32,n=12,2,0,7 | -39.8 [-68.6 to 93.3] | -92.2 [-96.1 to -88.2] |  | -73.5 [-91.8 to 47.0]
  Naive CD19+CD20+CD27-,Week 40,n=13,2,0,7: number analyzed (Participants) | 13 | 2 | 0 | 7
  Naive CD19+CD20+CD27-,Week 40,n=13,2,0,7 | -6.8 [-56.0 to 208.6] | -92.6 [-96.9 to -88.2] |  | -68.4 [-91.2 to 10.6]
  Naive CD19+CD20+CD27-,Week 52,n=13,2,0,6: number analyzed (Participants) | 13 | 2 | 0 | 6
  Naive CD19+CD20+CD27-,Week 52,n=13,2,0,6 | 17.1 [-36.8 to 104.9] | -92.7 [-95.2 to -90.2] |  | -77.9 [-94.3 to 13.6]
  Plasma CD19+CD20-CD138+,Day0,n=11,2,8,0: number analyzed (Participants) | 11 | 2 | 8 | 0
  Plasma CD19+CD20-CD138+,Day0,n=11,2,8,0 | -96.2 [-100.0 to -75.6] | 45.8 [-98.7 to 190.3] | -56.7 [-78.4 to 19.8] |
  Plasma CD19+CD20-CD138+,Week8,n=10,2,7,0: number analyzed (Participants) | 10 | 2 | 7 | 0
  Plasma CD19+CD20-CD138+,Week8,n=10,2,7,0 | -100.0 [-100.0 to -98.3] | 752.7 [-96.0 to 1601.4] | -88.6 [-92.3 to -44.5] |
  Plasma CD19+CD20-CD138+, Week16,n=9,2,7,0: number analyzed (Participants) | 9 | 2 | 7 | 0
  Plasma CD19+CD20-CD138+, Week16,n=9,2,7,0 | -97.8 [-99.3 to -96.5] | 535.2 [-90.7 to 1161.1] | -53.5 [-95.0 to -37.8] |
  Plasma CD19+CD20-CD138+,Week24,n=9,2,7,0: number analyzed (Participants) | 9 | 2 | 7 | 0
  Plasma CD19+CD20-CD138+,Week24,n=9,2,7,0 | -88.8 [-99.6 to -74.3] | 68.9 [-95.5 to 233.3] | -79.1 [-88.6 to 844.5] |
  Plasma CD19+CD20-CD138+,Week32,n=9,2,0,7: number analyzed (Participants) | 9 | 2 | 0 | 7
  Plasma CD19+CD20-CD138+,Week32,n=9,2,0,7 | -76.0 [-85.9 to -34.1] | 182.5 [-99.0 to 463.9] |  | -41.3 [-93.7 to 87.3]
  Plasma CD19+CD20-CD138+,Week40,n=9,2,0,7: number analyzed (Participants) | 9 | 2 | 0 | 7
  Plasma CD19+CD20-CD138+,Week40,n=9,2,0,7 | -53.4 [-80.9 to -13.2] | -9.0 [-100.0 to 81.9] |  | -86.5 [-95.7 to 362.8]
  Plasma CD19+CD20-CD138+,Week52,n=9,2,0,6: number analyzed (Participants) | 9 | 2 | 0 | 6
  Plasma CD19+CD20-CD138+,Week52,n=9,2,0,6 | -75.5 [-93.7 to -37.9] | -43.8 [-100.0 to 12.5] |  | -53.8 [-91.1 to 60.4]
  Plasmacytoid CD19+CD20+CD138+,Day 0,n=11,2,8,0: number analyzed (Participants) | 11 | 2 | 8 | 0
  Plasmacytoid CD19+CD20+CD138+,Day 0,n=11,2,8,0 | -98.9 [-99.7 to -94.7] | 118.1 [-85.6 to 321.9] | -75.5 [-96.5 to -25.0] |
  Plasmacytoid CD19+CD20+CD138+,Week8,n=10,2,7,0: number analyzed (Participants) | 10 | 2 | 7 | 0
  Plasmacytoid CD19+CD20+CD138+,Week8,n=10,2,7,0 | -97.6 [-99.8 to -94.6] | 14.1 [-90.6 to 118.8] | -75.0 [-98.2 to 54.9] |
  Plasmacytoid CD19+CD20+CD138+,Week16,n=9,2,7,0: number analyzed (Participants) | 9 | 2 | 7 | 0
  Plasmacytoid CD19+CD20+CD138+,Week16,n=9,2,7,0 | -98.7 [-100.0 to -96.8] | 226.3 [-94.4 to 546.9] | -75.9 [-95.5 to 526.4] |
  Plasmacytoid CD19+CD20+CD138+,Week24,n=9,2,7,0: number analyzed (Participants) | 9 | 2 | 7 | 0
  Plasmacytoid CD19+CD20+CD138+,Week24,n=9,2,7,0 | -98.5 [-98.8 to -93.0] | -16.3 [-95.0 to 62.5] | -15.0 [-65.0 to 254.7] |
  Plasmacytoid CD19+CD20+CD138+,Week32,n=9,2,0,7: number analyzed (Participants) | 9 | 2 | 0 | 7
  Plasmacytoid CD19+CD20+CD138+,Week32,n=9,2,0,7 | -95.4 [-97.9 to -82.2] | -24.1 [-85.6 to 37.5] |  | -52.5 [-96.3 to 728.3]
  Plasmacytoid CD19+CD20+CD138+,Week40,n=9,2,0,7: number analyzed (Participants) | 9 | 2 | 0 | 7
  Plasmacytoid CD19+CD20+CD138+,Week40,n=9,2,0,7 | -93.4 [-94.4 to -41.4] | -31.3 [-100.0 to 37.5] |  | 2.5 [-94.0 to 52.8]
  Plasmacytoid CD19+CD20+CD138+,Week 52,n=9,2,0,6: number analyzed (Participants) | 9 | 2 | 0 | 6
  Plasmacytoid CD19+CD20+CD138+,Week 52,n=9,2,0,6 | -96.1 [-98.5 to -73.9] | 202.5 [-91.9 to 496.9] |  | 32.2 [10.0 to 69.8]
  SLE Subset CD19+CD38b+CD27b+Lymph,Day0,n=11,2,8,0: number analyzed (Participants) | 11 | 2 | 8 | 0
  SLE Subset CD19+CD38b+CD27b+Lymph,Day0,n=11,2,8,0 | -28.3 [-60.4 to 43.8] | -67.9 [-93.2 to -42.6] | -66.7 [-78.1 to 215.2] |
  SLE Subset CD19+CD38b+CD27b+Lymph,Week8,n=10,2,7,0: number analyzed (Participants) | 10 | 2 | 7 | 0
  SLE Subset CD19+CD38b+CD27b+Lymph,Week8,n=10,2,7,0 | -30.5 [-52.0 to 137.2] | -91.7 [-96.6 to -86.7] | -71.9 [-89.0 to 121.3] |
  SLE Subset CD19+CD38b+CD27b+Lymph,Week16,n=9,2,7,0: number analyzed (Participants) | 9 | 2 | 7 | 0
  SLE Subset CD19+CD38b+CD27b+Lymph,Week16,n=9,2,7,0 | 21.3 [-82.6 to 157.5] | -74.2 [-97.0 to -51.3] | -48.6 [-82.1 to 204.4] |
  SLE Subset CD19+CD38b+CD27b+Lymph,Week24,n=9,2,7,0: number analyzed (Participants) | 9 | 2 | 7 | 0
  SLE Subset CD19+CD38b+CD27b+Lymph,Week24,n=9,2,7,0 | 25.2 [-48.1 to 168.6] | -64.7 [-75.1 to -54.2] | 152.3 [18.0 to 485.1] |
  SLE Subset CD19+CD38b+CD27b+Lymph,Week32,n=9,2,0,7: number analyzed (Participants) | 9 | 2 | 0 | 7
  SLE Subset CD19+CD38b+CD27b+Lymph,Week32,n=9,2,0,7 | -8.4 [-75.9 to 135.1] | -37.5 [-82.8 to 7.8] |  | -4.6 [-93.8 to 305.8]
  SLE Subset CD19+CD38b+CD27b+Lymph,Week40,n=9,2,0,7: number analyzed (Participants) | 9 | 2 | 0 | 7
  SLE Subset CD19+CD38b+CD27b+Lymph,Week40,n=9,2,0,7 | -8.5 [-24.5 to 87.2] | -66.3 [-90.6 to -42.1] |  | -24.6 [-85.3 to 450.6]
  SLE Subset CD19+CD38b+CD27b+Lymph,Week52,n=9,2,0,6: number analyzed (Participants) | 9 | 2 | 0 | 6
  SLE Subset CD19+CD38b+CD27b+Lymph,Week52,n=9,2,0,6 | -23.5 [-54.0 to 20.1] | -81.4 [-85.9 to -77.0] |  | 0.7 [-40.8 to 383.0]
  CD20+ Day 0,n=16,2,8,0: number analyzed (Participants) | 16 | 2 | 8 | 0
  CD20+ Day 0,n=16,2,8,0 | -75.2 [-89.1 to -58.7] | -88.1 [-95.8 to -80.5] | -77.1 [-86.8 to -22.0] |
  CD20+ Week 8,n=15,2,5,0: number analyzed (Participants) | 15 | 2 | 5 | 0
  CD20+ Week 8,n=15,2,5,0 | -79.9 [-89.1 to -58.0] | -91.0 [-95.8 to -86.2] | -80.9 [-81.5 to -11.1] |
  CD20+,Week16,n=14,2,6,0: number analyzed (Participants) | 14 | 2 | 6 | 0
  CD20+,Week16,n=14,2,6,0 | -75.4 [-90.5 to -58.7] | -84.3 [-96.2 to -72.4] | -80.4 [-90.8 to -9.7] |
  CD20+,Week24,n=13,2,6,0: number analyzed (Participants) | 13 | 2 | 6 | 0
  CD20+,Week24,n=13,2,6,0 | -52.0 [-90.9 to 26.3] | -87.7 [-93.7 to -81.6] | -53.4 [-71.3 to 31.9] |
  CD20+,Week32,n=12,2,0,7: number analyzed (Participants) | 12 | 2 | 0 | 7
  CD20+,Week32,n=12,2,0,7 | -49.0 [-74.1 to 62.4] | -87.4 [-95.4 to -79.3] |  | -66.2 [-90.1 to 54.2]
  CD20+,Week40,n=13,2,0,7: number analyzed (Participants) | 13 | 2 | 0 | 7
  CD20+,Week40,n=13,2,0,7 | -15.2 [-60.0 to 145.6] | -86.6 [-96.2 to -77.0] |  | -59.1 [-88.7 to 16.7]
  CD20+,Week52,n=13,2,0,6: number analyzed (Participants) | 13 | 2 | 0 | 6
  CD20+,Week52,n=13,2,0,6 | -12.0 [-45.0 to 88.1] | -89.8 [-94.6 to -85.1] |  | -71.8 [-92.7 to 19.4]
  Activated CD19+CD20+CD69+,Day0, n=11,1,8,0: number analyzed (Participants) | 11 | 1 | 8 | 0
  Activated CD19+CD20+CD69+,Day0, n=11,1,8,0 | -99.8 [-100.0 to -91.7] | -86.1 [-86.1 to -86.1] | -65.1 [-93.6 to -2.1] |
  Activated CD19+CD20+CD69+, Week8, n=10,1,7,0: number analyzed (Participants) | 10 | 1 | 7 | 0
  Activated CD19+CD20+CD69+, Week8, n=10,1,7,0 | -99.6 [-100.0 to -98.2] | -97.1 [-97.1 to -97.1] | -76.3 [-100.0 to 2141.7] |
  Activated CD19+CD20+CD69+, Week16, n=9,1,7,0: number analyzed (Participants) | 9 | 1 | 7 | 0
  Activated CD19+CD20+CD69+, Week16, n=9,1,7,0 | -98.9 [-99.4 to -98.3] | -93.4 [-93.4 to -93.4] | -72.3 [-98.9 to -22.9] |
  Activated CD19+CD20+CD69+,Week24, n=9,1,7,0: number analyzed (Participants) | 9 | 1 | 7 | 0
  Activated CD19+CD20+CD69+,Week24, n=9,1,7,0 | -99.7 [-100.0 to -95.3] | -94.2 [-94.2 to -94.2] | -50.9 [-95.6 to 80.0] |
  Activated CD19+CD20+CD69+,Week32, n=9,1,0,7: number analyzed (Participants) | 9 | 1 | 0 | 7
  Activated CD19+CD20+CD69+,Week32, n=9,1,0,7 | -98.0 [-99.8 to -97.4] | -86.9 [-86.9 to -86.9] |  | -54.5 [-74.1 to 975.0]
  Activated CD19+CD20+CD69+, Week40, n=9,1,0,7: number analyzed (Participants) | 9 | 1 | 0 | 7
  Activated CD19+CD20+CD69+, Week40, n=9,1,0,7 | -98.1 [-99.8 to -96.7] | -100.0 [-100.0 to -100.0] |  | -47.5 [-100.0 to -24.6]
  Activated CD19+CD20+CD69+, Week52, n=9,1,0,6: number analyzed (Participants) | 9 | 1 | 0 | 6
  Activated CD19+CD20+CD69+, Week52, n=9,1,0,6 | -96.9 [-99.3 to -93.6] | -100.0 [-100.0 to -100.0] |  | -27.4 [-57.5 to 50.0]

11. Secondary Outcome: Percentage Change From 24 Week in B Cell Subsets: Treatment Holiday Group (Re-start Phase)
Description: Blood samples were collected at indicated time-points for analysis of Activated B cells subsets like Activated CD19+CD20+CD69+, CD20+, Memory CD19+CD20+CD27+, Naive CD19+CD20+CD27-, Plasma CD19+CD20-CD138+, Plasmacytoid CD19+CD20+CD138+, and SLE Subset CD19+CD38b+CD27b+Lymph. Percentage change from Week 24 of present study was calculated as 100*(value at specified visit - Week 24 value) divided by week 24 value. The data below is only reported for the Treatment Holiday Group (Re-start phase). Participants in this group restarted belimumab therapy one day after Week 24, hence the Baseline for this outcome measure was Week 24 visit. No other groups were measured for this outcome.
Time Frame: Week 24, 32, 40 and 52 weeks
Population: ITT Population. Participants in this group restarted belimumab therapy one day after Week 24, hence the Baseline for this outcome measure was Week 24 visit. The data below is only reported for the Treatment Holiday Group and no other groups were measured.
Measure: Median (Inter-Quartile Range); unit: Percent change
Arm/Group | Treatment Holiday Group - Re-start Phase
Number analyzed (Participants) | 11
Percent change
  Memory CD19+CD20+CD27+, Week 32: number analyzed (Participants) | 8
  Memory CD19+CD20+CD27+, Week 32 | 100.0 [40.5 to 250.0]
  Memory CD19+CD20+CD27+, Week 40: number analyzed (Participants) | 9
  Memory CD19+CD20+CD27+, Week 40 | 83.3 [48.3 to 366.7]
  Memory CD19+CD20+CD27+,Week52: number analyzed (Participants) | 8
  Memory CD19+CD20+CD27+,Week52 | 66.7 [12.4 to 233.3]
  Naive CD19+CD20+CD27-,Week 32: number analyzed (Participants) | 8
  Naive CD19+CD20+CD27-,Week 32 | -19.0 [-58.8 to 31.1]
  Naive CD19+CD20+CD27-,Week 40: number analyzed (Participants) | 9
  Naive CD19+CD20+CD27-,Week 40 | -12.5 [-61.8 to 7.7]
  Naive CD19+CD20+CD27-,Week52: number analyzed (Participants) | 8
  Naive CD19+CD20+CD27-,Week52 | -35.6 [-84.8 to -7.9]
  Plasma CD19+CD20-CD138+,Week32: number analyzed (Participants) | 10
  Plasma CD19+CD20-CD138+,Week32 | -16.3 [-71.4 to 237.8]
  Plasma CD19+CD20-CD138+, Week40 | -59.8 [-73.7 to 18.5]
  Plasma CD19+CD20-CD138+,Week52: number analyzed (Participants) | 10
  Plasma CD19+CD20-CD138+,Week52 | -48.0 [-92.4 to 188.9]
  Plasmacytoid CD19+CD20+CD138+,Week32: number analyzed (Participants) | 9
  Plasmacytoid CD19+CD20+CD138+,Week32 | -35.7 [-69.3 to 133.5]
  Plasmacytoid CD19+CD20+CD138+,Week40: number analyzed (Participants) | 10
  Plasmacytoid CD19+CD20+CD138+,Week40 | -64.3 [-89.4 to -56.9]
  Plasmacytoid CD19+CD20+CD138+,Week52: number analyzed (Participants) | 9
  Plasmacytoid CD19+CD20+CD138+,Week52 | -55.0 [-72.7 to -52.1]
  SLE SubsetCD19+CD38b+CD27b+Lymph,Week32: number analyzed (Participants) | 10
  SLE SubsetCD19+CD38b+CD27b+Lymph,Week32 | -55.4 [-71.6 to -27.2]
  SLE SubsetCD19+CD38b+CD27b+Lymph,Week40 | -56.9 [-75.3 to -0.7]
  SLE SubsetCD19+CD38b+CD27b+Lymph,Week52: number analyzed (Participants) | 10
  SLE SubsetCD19+CD38b+CD27b+Lymph,Week52 | -67.2 [-79.7 to -41.0]
  CD20+, Week 32: number analyzed (Participants) | 8
  CD20+, Week 32 | -3.3 [-45.2 to 29.7]
  CD20+, Week 40: number analyzed (Participants) | 9
  CD20+, Week 40 | 2.2 [-51.4 to 17.4]
  CD20+, Week 52: number analyzed (Participants) | 8
  CD20+, Week 52 | -20.0 [-78.9 to 30.8]
  Activated CD19+CD20+CD69+,Week32: number analyzed (Participants) | 9
  Activated CD19+CD20+CD69+,Week32 | -28.8 [-75.8 to 64.7]
  Activated CD19+CD20+CD69+,Week40: number analyzed (Participants) | 10
  Activated CD19+CD20+CD69+,Week40 | -23.8 [-88.1 to 191.2]
  Activated CD19+CD20+CD69+,Week52: number analyzed (Participants) | 9
  Activated CD19+CD20+CD69+,Week52 | -66.7 [-89.0 to 87.7]

12. Secondary Outcome: SELENA SLEDAI Scores Change From Baseline
Description: SELENA SLEDAI assessments consist of 24 individual weighted items in which signs and symptoms, laboratory tests, and physician's assessment for each of 9 organ systems are given a weighted score and summed if present (marked 'Yes') at the time of the visit or in the preceding 10 days. The maximum theoretical score is 105 (all 24 descriptors present simultaneously) with 0 indicating inactive disease (marked 'No'). Data are reported at the specified time-points from Day 0 (of present study) up to Week 52. Baseline is defined as the Day 0 from parent studies. Change from Baseline is equal to (Value at specified visit minus Baseline value).
Time Frame: Baseline (Day 0 from parent studies); Day 0 and 4, 8, 12, 16, 20, 24, 28, 32,36, 40, 44, 48 and 52 weeks
Population: ITT Population. Only those participants with data available at the specified time points were analyzed (represented by n= X in the category titles).
Measure: Mean (Standard Deviation); unit: Scores on a scale
Groups:
- Long-term Discontinuation: Participants in this group discontinued belimumab 10 mg/kg therapy for 52 weeks but remained on standard of care therapy. Participants from BEL114333 (NCT01597622), BEL112233 (NCT00724867) and BEL112626 (NCT00583362) were part of this group. Participants had been treated with belimumab for at least 6 months in one of these continuation studies but had withdrawn from belimumab therapy for no longer than 8 weeks prior to entry into this study.
Arm/Group | Long-term Discontinuation | Treatment Control Group | Treatment Holiday Group - Holiday Phase | Treatment Holiday Group - Re-start Phase
Number analyzed (Participants) | 39 | 29 | 12 | 11
Scores on a scale
  Day 0,n=39,29,12, 0: number analyzed (Participants) | 39 | 29 | 12 | 0
  Day 0,n=39,29,12, 0 | -6.2 (4.12) | -6.9 (3.62) | -6.3 (4.31) |
  Week 4,n=39,29,12, 0: number analyzed (Participants) | 39 | 29 | 12 | 0
  Week 4,n=39,29,12, 0 | -5.9 (5.07) | -6.6 (3.44) | -6.1 (4.01) |
  Week 8,n=38,29, 11,0: number analyzed (Participants) | 38 | 29 | 11 | 0
  Week 8,n=38,29, 11,0 | -6.4 (4.18) | -7.0 (3.73) | -5.9 (4.16) |
  Week 12,n=38,29, 11,0: number analyzed (Participants) | 38 | 29 | 11 | 0
  Week 12,n=38,29, 11,0 | -6.1 (4.28) | -7.0 (3.75) | -6.3 (3.95) |
  Week 16,n=36,27, 11,0: number analyzed (Participants) | 36 | 27 | 11 | 0
  Week 16,n=36,27, 11,0 | -6.4 (5.21) | -6.8 (4.05) | -6.1 (3.96) |
  Week 20,n=36,27, 11,0: number analyzed (Participants) | 36 | 27 | 11 | 0
  Week 20,n=36,27, 11,0 | -6.9 (4.17) | -6.9 (3.23) | -6.1 (3.96) |
  Week 24,n=36,27, 11,0: number analyzed (Participants) | 36 | 27 | 11 | 0
  Week 24,n=36,27, 11,0 | -6.4 (4.45) | -6.7 (3.45) | -5.4 (4.01) |
  Week 28,n=35,27,0,10: number analyzed (Participants) | 35 | 27 | 0 | 10
  Week 28,n=35,27,0,10 | -5.8 (4.22) | -7.0 (3.32) |  | -5.5 (5.36)
  Week 32,n=34,27,0,11: number analyzed (Participants) | 34 | 27 | 0 | 11
  Week 32,n=34,27,0,11 | -5.7 (4.59) | -7.1 (3.38) |  | -6.1 (4.01)
  Week 36,n=34,27,0,11: number analyzed (Participants) | 34 | 27 | 0 | 11
  Week 36,n=34,27,0,11 | -5.0 (4.42) | -6.7 (3.59) |  | -5.9 (4.01)
  Week 40,n=34,27,0,11: number analyzed (Participants) | 34 | 27 | 0 | 11
  Week 40,n=34,27,0,11 | -5.2 (4.30) | -7.2 (3.37) |  | -6.6 (4.30)
  Week 44,n=34,27,0,11: number analyzed (Participants) | 34 | 27 | 0 | 11
  Week 44,n=34,27,0,11 | -5.8 (4.15) | -7.3 (3.49) |  | -6.3 (4.65)
  Week 48,n=33,27,0,11: number analyzed (Participants) | 33 | 27 | 0 | 11
  Week 48,n=33,27,0,11 | -5.7 (4.30) | -7.3 (3.28) |  | -6.1 (3.91)
  Week 52,n=33,27,0,11: number analyzed (Participants) | 33 | 27 | 0 | 11
  Week 52,n=33,27,0,11 | -5.0 (4.39) | -6.9 (3.69) |  | -5.5 (4.08)

13. Secondary Outcome: Number of Days of Daily Prednisone Dose >=7.5 mg/Day and/or Increased by 25 Percent From Day 0 of This Study
Description: All corticosteroids are converted to a prednisone equivalent average daily dose (mg/day). The average daily dose at Day 0 was used to assess the relative change in daily dose on a given day. The average daily dose at Day 0 was calculated as sum of the daily dose across all days from the Screening visit date up to and including Day 0 visit date divided by the number of days in the time period. Data reported are the median number of days on which the specified criteria was met for Day 0 to Week 24, Week 24 to Week 52, Day 0 to Week 52. For treatment holiday group, Day 0 to Week 24 corresponds to holiday phase, Week 24 to Week 52 corresponds to treatment Re-start phase.
Time Frame: Day 0 to Week 24; Week 24 to Week 52; Day 0 to Week 52
Population: ITT Population. Only those participants who met specified criteria (>=7.5 mg/day and/or increased by 25%) within specified time period were analyzed (represented by n= X in the category titles).
Measure: Median (Full Range); unit: Days
Arm/Group | Long-term Discontinuation Group | Treatment Control Group | Treatment Holiday Group
Number analyzed (Participants) | 13 | 12 | 6
Days
  Day 0 to Week 24, n=11, 12, 6: number analyzed (Participants) | 11 | 12 | 6
  Day 0 to Week 24, n=11, 12, 6 | 143.0 [3 to 173] | 170.0 [67 to 175] | 168.0 [61 to 170]
  Day 0 to Week 52, n=13, 12, 6 | 278.0 [5 to 369] | 364.0 [145 to 392] | 364.0 [250 to 366]
  Week 24 to Week 52, n=10, 9, 5: number analyzed (Participants) | 10 | 9 | 5
  Week 24 to Week 52, n=10, 9, 5 | 167.5 [1 to 201] | 196.0 [189 to 217] | 196.0 [194 to 196]

14. Secondary Outcome: Number of Days of Daily Prednisone Dose <=7.5 mg/Day and/or Decreased by 25 Percent From Day 0 of This Study
Description: as for outcome 13
Time Frame: Day 0 to Week 24; Week 24 to Week 52; Day 0 to Week 52
Population: ITT Population. Only those participants who met specified criteria (<=7.5 mg/day and/or decreased by 25%) within specified time period were analyzed (represented by n= X in the category titles).
Measure: Median (Full Range); unit: Days
Arm/Group | Long-term Discontinuation Group | Treatment Control Group | Treatment Holiday Group
Number analyzed (Participants) | 25 | 19 | 6
Days
  Day 0 to Week 24, n=23,19, 6: number analyzed (Participants) | 23 | 19 | 6
  Day 0 to Week 24, n=23,19, 6 | 168.0 [23 to 181] | 168.0 [26 to 175] | 166.0 [49 to 170]
  Day 0 to Week 52, n=25,19, 6 | 362.0 [23 to 385] | 364.0 [91 to 391] | 364.0 [49 to 370]
  Week 24 to Week 52, n=24,18, 5: number analyzed (Participants) | 24 | 18 | 5
  Week 24 to Week 52, n=24,18, 5 | 195.0 [1 to 208] | 196.0 [189 to 225] | 200.0 [189 to 203]

ADVERSE EVENTS:
Time Frame: Non-serious adverse events and serious adverse events (SAE) were collected up to 52 weeks for all treatment groups. For Treatment Control and Treatment Holiday Re-start, it also included 16 weeks follow up after the last dose of belimumab for participants who did not continue in Maintenance phase. For Maintenance phase, non-SAE and SAE were collected until Week 48 of subsequent years (Maintenance is Year 2, 3, 4) and includes 16 weeks follow up after last dose of belimumab.
Description: Treatment holiday group had two phases holiday phase was Day 0 visit to Week 24/Treatment Re-start phase and Re-start phase started one day after Week 24 up to Week 52. Non-serious adverse events and SAEs were collected for ITT Population.
Groups:
- Treatment Phase: Long-term Discontinuation Group: Participants in this group discontinued belimumab 10 mg/kg therapy for 52 weeks but remained on standard of care therapy. Participants from BEL114333 (NCT01597622), BEL112233 (NCT00724867) and BEL112626 (NCT00583362) were part of this group. Participants had been treated with belimumab for at least 6 months in one of these continuation studies but had withdrawn from belimumab therapy for no longer than 8 weeks prior to entry into this study.
- Treatment Phase: Treatment Control Group: Participants in this group continued to receive monthly belimumab 10 mg/kg therapy, in addition to standard of care SLE therapy for 52 weeks. Participants from BEL113750 (NCT01345253) and BEL114333 (NCT01597622) were part of this group. Participants had been treated with belimumab for at least 6 months in one of these continuation studies prior to entry into this study. Eligible participants on completion of 52-weeks entered Maintenance period and received belimumab 10 mg/kg every 4 weeks until Week 48 of subsequent years (Maintenance is Year 2, 3, 4).
- Treatment Phase: Treatment Holiday Group - Holiday Phase: Participants in the Treatment Holiday Group underwent a 24-week belimumab treatment holiday while remaining on standard of care SLE therapy, Holiday Phase was Day 0 visit to Week 24/Treatment Re-start phase. Participants from BEL113750 (NCT01345253) and BEL114333 (NCT01597622) were part of this group. Participants had been treated with belimumab for at least 6 months in one of these continuation studies prior to entry into this study. In the event of a severe flare, participants were allowed to enter Maintenance Phase and receive belimumab 10 mg/Kg every 4 weeks until Week 48 of subsequent years (Maintenance is Year 2, 3, 4).
- Treatment Phase: Treatment Holiday Group - Re-start Phase: Following Treatment holiday phase for 24 weeks, participants re-started belimumab therapy for 28 weeks while receiving standard of care SLE therapy for 52 weeks. Re-start Phase started one day after Week 24 up to Week 52. Participants from BEL113750 (NCT01345253) and BEL114333 (NCT01597622) were part of this group. Participants had been treated with belimumab for at least 6 months in one of these continuation studies prior to entry into this study. Eligible participants on completion of 52-weeks entered Maintenance period and received belimumab 10 mg/kg every 4 weeks until Week 48 of subsequent years (Maintenance is Year 2, 3, 4).
- Maintenance Phase: Treatment Control; Maintenance Phase: Treatment Holiday: Participants from BEL113750 (NCT01345253) and BEL114333 (NCT01597622) were part of this group. Eligible participants on completion of 52-weeks entered Maintenance period and received belimumab 10 mg/kg every 4 weeks until Week 48 of subsequent years (Maintenance is Year 2, 3, 4).
Arm/Group | Treatment Phase: Long-term Discontinuation Group | Treatment Phase: Treatment Control Group | Treatment Phase: Treatment Holiday Group - Holiday Phase | Treatment Phase: Treatment Holiday Group - Re-start Phase | Maintenance Phase: Treatment Control | Maintenance Phase: Treatment Holiday
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/29 | 0/12 | 0/11 | 0/16 | 0/10
Serious Adverse Events (participants affected / at risk) | 6/39 | 2/29 | 0/12 | 1/11 | 0/16 | 0/10
Other Adverse Events (participants affected / at risk) | 30/39 | 18/29 | 7/12 | 9/11 | 4/16 | 8/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Phase: Long-term Discontinuation Group (N=39) | Treatment Phase: Treatment Control Group (N=29) | Treatment Phase: Treatment Holiday Group - Holiday Phase (N=12) | Treatment Phase: Treatment Holiday Group - Re-start Phase (N=11) | Maintenance Phase: Treatment Control (N=16) | Maintenance Phase: Treatment Holiday (N=10)
Diarrhoea infectious (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia pseudomonal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lupus nephritis (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pericarditis lupus (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Generalised oedema (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Phase: Long-term Discontinuation Group (N=39) | Treatment Phase: Treatment Control Group (N=29) | Treatment Phase: Treatment Holiday Group - Holiday Phase (N=12) | Treatment Phase: Treatment Holiday Group - Re-start Phase (N=11) | Maintenance Phase: Treatment Control (N=16) | Maintenance Phase: Treatment Holiday (N=10)
Nasopharyngitis (Infections and infestations) | 10 (16) | 5 (16) | 1 (2) | 4 (4) | 2 (5) | 4 (7)
Upper respiratory tract infection (Infections and infestations) | 5 (5) | 2 (4) | 2 (4) | 1 (1) | 2 (2) | 1 (1)
Sinusitis (Infections and infestations) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection bacterial (Infections and infestations) | 3 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Cystitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (3)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Otitis externa bacterial (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tinea versicolour (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (10) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 4 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (8) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 3 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dental caries (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Periodontal disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Increased tendency to bruise (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 4 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deafness (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chalazion (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ocular discomfort (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Angular cheilitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Viral myositis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gingivitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myopathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intervertebral disc displacement (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Polymyositis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chillblains (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Benign neoplasm of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Drug eruption (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Study limitations include the small sample size and differences in Day 0 characteristics between Long-term Discontinuation and Treatment Control groups, which limits the ability to draw inferences.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Statistical Analysis Plan (2019-01-30): https://cdn.clinicaltrials.gov/large-docs/56/NCT02119156/SAP_000.pdf
  • Study Protocol (2017-09-12): https://cdn.clinicaltrials.gov/large-docs/56/NCT02119156/Prot_001.pdf